CLINICAL TRIAL: NCT05124756
Title: Effects of Bioelectric Stimulation on Kidney Function and Sarcopenia in Patients With Non-Dialysis Dependent Chronic Kidney Disease (CKD): Randomized Controlled Trial
Brief Title: Effects of Bioelectric Stimulation in Patients With Non-Dialysis Dependent Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Leonhardt Ventures LLC (Industry); Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CKD_EE_Klotho
Record Dates: First submitted 2021-10-15; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Renal Insufficiency, Chronic; Electric Stimulation
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioelectric stimulation (Experimental): Bioelectric stimulation on quadriceps muscle and kidneys: 45 minutes, 3 times/week, 8 weeks, 24 sessions.
  Interventions: Device: Bioelectric stimulation
- Control (No Intervention): No intervention.

INTERVENTIONS:
Device: Bioelectric stimulation — The sessions will include 20 minutes for stimulation of the thigh muscles and 45 minutes for stimulation of the kidneys. The electrodes will be placed on the motor point of the quadriceps muscle in both lower limbs. The neuromuscular electric stimulation will be applied by symmetrical biphasic pulsed current, at an 80 Hz frequency, 400 ms pulse width, 10 s contraction time, rest time decreasing as the protocol advanced, at reciprocal mode. The intensity will be individually adjusted to produce visible muscle contraction. Concomitant, two electrodes will be placed in the abdominal corresponding to the kidney anatomical site and two electrodes on the dorsal region at the level of the 10th thoracic vertebra. The stimulation of the kidneys will include in addition to Klotho, precise signals for several pro-regenerative proteins. The intensity of the electric current will be individually adjusted to sensory stimulation.
  Arms: Bioelectric stimulation

SUMMARY:
Chronic kidney disease (CKD) consists of kidney damage, with a consequent progressive and irreversible loss of kidney function. In the early stages of the disease, there is already a reduction in circulating levels of α-klotho protein, which is related to worsening renal function. Therapeutic strategies that increase serum α-klotho levels can be of great value in the treatment of CKD. Electrical stimulation contributes to the reduction of reactive oxygen species, DNA damage and improves the efficiency rate of dialysis, suggesting a systemic effect in patients with end-stage CKD. The aim of this study is to evaluate the effects of bioelectric stimulation on renal function and physical capacity in patients with CKD. For this, patients will be randomized into bioelectric stimulation or a control group. Bioelectric stimulation will be performed three times a week for eight weeks. The control group will only be evaluated and re-evaluated. The following pre-and post-intervention assessments will be performed: analysis of the plasma content of α-Klotho and soluble creatinine to assess renal function, six-minute walk test to assess functional capacity; dosage of interleukins and tumor necrosis factor to analyze the inflammatory profile; sit and stand test with 10 repetitions and load cell dynamometry to assess lower limb muscle strength and application of the EuroQoL-5D questionnaire for quality of life. Biochemical analyzes for renal function and inflammatory profile will also be performed after four weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years of age;
* CKD with glomerular filtration rate (GFR) between 15-59 ml/min (III and IV stage of CKD) for more than 3 months;
* To be able to ambulate > 300 meters in 6 minutes walk test.

Exclusion Criteria:

* Cognitive dysfunction that prevents the performance of evaluations, as well as an inability to understand and sign the informed consent form;
* Intolerance to the electrostimulator and/or alteration of skin sensitivity;
* Skin lesions/burns at the electrode placement site;
* Patients with stroke in past 6 months with residual limitation to ambulation;
* Disabling musculoskeletal disease;
* Uncontrolled hypertension (systolic blood pressure > 230 mmHg and diastolic blood pressure > 120 mmHg);
* Grade III or IV heart failure (NYHA);
* Patient with a pacemaker;
* Uncontrolled diabetes (fasting blood glucose > 250 mg/dL);
* Unstable angina;
* Coronary stent placement in past 3 months;
* Recent acute myocardial infarction (two months);
* Fever and/or infectious disease;
* Peripheral vascular disease in the lower limbs that limits ambulation or deep vein thrombosis;
* Chronic obstructive lung disease that limits ambulation or need for oxygen therapy;
* Obesity (Body Mass Index≥35);
* Patient with active cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-25 (Estimated); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-10-25 (Estimated)

PRIMARY OUTCOMES:
Change from kidney function | Baseline, after 4 weeks and after 8 weeks
  The kidney function will be assessed through the blood collection and dosage of serum creatinine
Change from kidney function | Baseline, after 4 weeks and after 8 weeks
  The kidney function will be assessed through the blood collection and dosage of α-klotho protein expression
Change from kidney function | Baseline, after 4 weeks and after 8 weeks
  The kidney function will be assessed through the glomerular filtration rate

SECONDARY OUTCOMES:
Change in functional capacity | Baseline and after 8 weeks
  Functional capacity will be assessed by change in distance covered in the six minute walk test
Change in muscle strength | Baseline and after 8 weeks
  Muscle strength will be evaluated by dynamometry by a load cell
Change in muscle strength of the lower limbs | Baseline and after 8 weeks
  Muscle strength of the lower limbs will be assessed by sit-and-stand test of 10 repetitions
Change in quality of life evaluation | Baseline and after 8 weeks
  The quality of life will be assessed by questionnaire EuroQol-5D health questionnaire
Adverse effects | After 8 weeks
  Adverse effects will be recorded in number of cases and type of event
Change in inflammatory profile | Baseline, after 4 weeks and after 8 weeks
  The inflammatory profile will be assessed through the blood collection and analysis of immunological marker interleukin 6
Change in inflammatory profile | Baseline, after 4 weeks and after 8 weeks
  The inflammatory profile will be assessed through the blood collection and analysis of immunological marker interleukin 10
Change in inflammatory profile | Baseline, after 4 weeks and after 8 weeks
  The inflammatory profile will be assessed through the blood collection and analysis of immunological marker tumor necrosis factor

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre

IPD SHARING:
Plan to Share IPD: No